CLINICAL TRIAL: NCT03892252
Title: Correlation Analysis of TCM Syndromes, TCM Constitution Types, Intestinal Microbial Evolution and Tumor Biological Characteristics in Colorectal Cancer Patients Before and After Surgery
Brief Title: Characteristics of Gut Microbiota in Patients With Colon Cancer of Different Traditional Chinese Medicine Syndromes
Status: Completed | Type: Observational
Sponsor: Wei Xu (Other)
Responsible Party: Sponsor-Investigator, Wei Xu, Professor, First Affiliated Hospital of Harbin Medical University
Organization: First Affiliated Hospital of Harbin Medical University (Other)
Other Study IDs: V1.0
Record Dates: First submitted 2019-03-14; First posted 2019-03-27 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Neoplasms
Keywords: gut microbiota; 16s rDNA sequebcing; TCM sydromes; TCM Constitution Types
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fecal
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- before surgery: no intervention(s)
  Interventions: Other: No intervention
- after surgery: no intervention(s)
  Interventions: Other: No intervention
- Normal colonoscopy: People who were diagnosed by colonoscopy without colorectal cancer.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Guided by the idea of combining disease differentiation with syndrome differentiation in traditional Chinese medicine, this study used the form of questionnaire to summarize the changes of TCM syndromes, TCM constitution types in colorectal cancer patients before and after surgery. The Next-generation sequencing technology was used to explore the changes and differences of intestinal microorganisms before and after surgery. The correlation between changes of TCM syndromes, TCM constitution types, intestinal microbial evolution and tumor biological characteristics in colorectal cancer patients before and after surgery was analyzed. To explore the rationality of TCM in the prevention and treatment of colorectal cancer recurrence and metastasis in order to guide the individualized treatment and dietary regulation of TCM.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative abdominal CT, colonoscopy and pathological examination were diagnosed as colorectal malignant tumor patients;
2. Having surgical indications;
3. Patients who were not treated with antibiotics or microbiological agents one week before surgery;
4. Patients who had not received radiotherapy and chemotherapy before surgery;
5. Patients or their legal representatives informed and agreed to participate in this clinical trial and signed a written informed consent;

Exclusion Criteria:

1. Have other cancer history;
2. Patients who have received invasive treatment within the past three months;
3. Inflammatory bowel disease such as ulcerative colitis or crohn's disease;
4. Combined with intestinal obstruction or intestinal perforation for emergency surgery;
5. Psychiatric history, can not join and standardize the completion of clinical investigators;
6. Pregnant or nursing women;
7. Patients treated with antibiotics or microbiological agents one week before surgery;
8. People have incomplete data;

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients admitted to the first affiliated hospital of Harbin medical university
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
According to the 16s rDNA sequencing results, characterize the intestinal microbiota characteristics of colon cancer patients with different TCM syndrome types and TCM constitutions before and after surgery | 2 year
According to the 16s rDNA sequencing results, analyze the differences in intestinal flora of colon cancer patients with different TCM syndromes and TCM constitutions before and after surgery and their correlations | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, Professor, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China